CLINICAL TRIAL: NCT01475318
Title: A Pilot Study on the Combined Use of Letrozole, Miferpristone and Misoprostol in Termination of First Trimester Pregnancy up to 63 Days Gestation
Brief Title: Study on Combined Use of Letrozole, Mifepristone and Misoprostol in Termination of Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mifemisolet
Record Dates: First submitted 2011-10-31; First posted 2011-11-21 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Complete Abortion
Keywords: complete abortion rate; side effects; induction-to-abortion interval
MeSH Terms: interventions — Mifepristone; Letrozole; Misoprostol

ARMS (1):
- misoprostol + mifepristone + letrozole (Experimental)
  Interventions: Drug: mifepristone; Drug: Letrozole; Drug: Misoprostol

INTERVENTIONS:
Drug: mifepristone — 200 mg mifepristone on day 1
Drug: Letrozole — Letrozole 10mg PO on day 1, day 2, and day 3
Drug: Misoprostol — misoprostol 800mcg PV on day 3

SUMMARY:
By using the combination of mifepristone (anti-progestin), misoprostol (progstanglandin which stimulates uterine contraction), and letrozole (aromatise inhibitor which reduces estrogen production), the abortion process will be more effective.

DETAILED DESCRIPTION:
After mifepristone was approved by the United States Food and Drug Administration in 2000, the combination of mifepristone 200 mg and vaginal use of misoprostol 800 mcg became almost a standard of care in early medical abortion up to 63 days of gestation. Misoprostol, a synthetic analogue of naturally occurring prostaglandin E1, has uterotonic effect and it can stimulate myometrial contraction and cause cervical ripening and dilatation. Progesterone maintains the uterus in a quiescent state by inducing hyperpolarization of the membrane of the myometrial cells and a greater change in electric potential is necessary before contractions can occur. Mifepristone is the anti-progestin that binds to the progesterone receptors and prevents endogenous progesterone from exerting is effects. It can also increase the sensitivity of the uterus to prostaglandins. The complete abortion rate achieved with this sequential regimen has been found to be up to 93-95%, which is higher than the rate achieved with either mifepristone or misoprostol alone.

Apart from progesterone, estrogen is another important hormone for the maintenance of pregnancy. Albrecht et al showed that 50% of the baboons miscarried when maternal estrogen synthesis was suppressed using aromatase inhibitors whereas all maintained their pregnancy when concomitant estradiol was given. Letrozole is a third-generation aromatase inhibitor which leads to reduced production of estrogen and has specific actions at clinical doses with no effect on basal levels of cortisol and aldosterone. Shi et al found that the combinations of anti-progestin with aromatase inhibitor act synergistically to induce 100% abortion rate in rats, with little effect of antiprogestin or aromatase inhibitor when administered alone. Lee et al conducted the first pilot study of the effect of letrozole on medical abortions of up to 9 weeks gestation in humans. When 7.5 mg letrozole was combined with 200 mg mifepristone, the abortion effect was not as great as those observed in animal study, with clinical complete abortion rate of 71% only. On the other hand, when 7.5 mg letrozole was given daily for 2 days followed by 800 mcg vaginal misoprostol, this regimen was associated with a clinical complete abortion rate of 80% and 87.5% with gestation of less than 63 days and gestation of less than 49 days respectively. Hormonal profiles revealed that letrozole led to significant reduction in oestradiol level, but progesterone level was not altered. The complete abortion rate achieved was noted to be higher when the dosage and duration of letrozole were increased to 10 mg for 3 days. There were no serious complications encountered in these 200 subjects, implying that these regimens are likely safe to use in humans.

Letrozole plays a role in medical termination through its principal effect on oestrodial synthesis, which is an important factor in the maintenance of early pregnancy. It is postulated that by combining both letrozole and mifepristone, together with misoprostol, a synergistic effect will be exerted as the depleted estrogen and progesterone level will be insufficient to support the pregnancy, and the uterotonic effect of misoprostol will hasten the abortion process, hence improving the complete abortion rate. The aim of this pilot study was to determine the complete abortion rate of vaginal misoprostol when given with mifepristone and letrozole for termination of first trimester pregnancy up to 9 weeks gestation.

ELIGIBILITY:
Inclusion Criteria:

* good general health
* older than the age of legal consent (i.e. >18 years old)
* requesting medical abortion and eligible for abortion
* on Day 1 of the study (day of letrozole and mifepristone administration) the duration of pregnancy not more than 63 days as confirmed by pelvic ultrasound examination
* intrauterine pregnancy (intrauterine amniotic sac seen in US)
* willing to use other than hormonal or intra-uterine contraception until the first menses after termination of pregnancy
* if treatment should fail agrees to termination of pregnancy with the surgical method
* willing and able to participate after the study has been explained
* haemoglobin higher than 10g/L, normal liver and renal function

Exclusion Criteria:

* a history or evidence of adrenal pathology, steroid-dependent cancer, porphyria, diastolic pressure over 95mm Hg, bronchial asthma, arterial hypotension
* a history or evidence of thrombo-embolism, severe or recurrent liver disease or pruritus of pregnancy
* the regular use of prescription drugs before admission to the study
* the presence of an IUCD in utero
* breast-feeding
* multiple pregnancies
* heavy smoker of more than 20 cigarettes per day
* any abnormal values in pre-treatment blood tests

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Complete abortion rate | from drug administration till return of next menses (average 4-6 weeks)
  If no suction evacuation is required before the return of next menstruation, it is classified as complete abortion

SECONDARY OUTCOMES:
the induction-to-abortion interval | drug administration to passage of abortus (average within 48 hours)
  The time between administration of misoprostol and spontaneous passage of tissue mass
incidence of side effects | drug administration (D1) till D43
  A list of side effects (nausea, vomiting, diarrhoea, fever, chills, headache, abdominal pain, bleeding) will be given to patient for record
the duration of bleeding | drug administration till cessation of bleeding (average 4-6 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Joyce Chai, Hong Kong, Hong Kong